CLINICAL TRIAL: NCT04437368
Title: EXPLORE: A Phase II, Outcomes Assessor-masked, Multicentre, Randomised Study to Evaluate the Safety and Efficacy of Two Doses of GT005 Administered as a Single Subretinal Injection in Subjects With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: EXPLORE: A Phase II Study to Evaluate the Safety and Efficacy of Two Doses of GT005
Acronym: EXPLORE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for interim analysis demonstrating futility (trial highly unlikely to meet efficacy outcome). The trial is not ending early because of medical problems or concerns.
Sponsor: Gyroscope Therapeutics Limited (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT005-02; CPPY988A12202 (Other: Novartis); 2019-003421-22 (EudraCT Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-18 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: Geographic atrophy; Retinal disease; Eye disease; Retinal degeneration; Macular atrophy; Dry age-related macular degeneration
MeSH Terms: conditions — Geographic Atrophy; Retinal Diseases; Eye Diseases; Retinal Degeneration; Anetoderma

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, outcomes assessor-masked multicentre, randomised study to evaluate the safety and efficacy of two doses of GT005 administered as a single subretinal injection in subjects with GA secondary to AMD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The overall objectives of the study are to evaluate the safety and efficacy (anatomical and functional visual outcomes) of two doses of GT005 in genetically defined subjects with GA due to AMD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GT005 Low dose [2E10 vg] (Experimental): GT005 Low dose [2E10 vg] (Parts 1 and 2)
  Interventions: Drug: GT005
- GT005 High dose [2E11 vg] (Experimental): GT005 High dose [2E11 vg] (Part 1)
  Interventions: Drug: GT005
- Untreated control (No Intervention): Untreated control (Parts 1 and 2)

INTERVENTIONS:
Drug: GT005 — GT005 is a recombinant, non-replicating AAV2 expressing human complement factor I (CFI). GT005 was administered as a single time subretinal injection into the study eye of subjects allocated to one of the two GT005 doses.
  Arms: GT005 High dose [2E11 vg]; GT005 Low dose [2E10 vg]

SUMMARY:
The purpose of this clinical study was to evaluate the safety and efficacy of two doses of GT005 administered as a single subretinal injection in subjects with geographic atrophy secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This was a Phase II, outcomes assessor-masked, multicentre, randomized study to assess the safety and efficacy of two doses of GT005 administered as a single-time subretinal injection in subjects with Geographic Atrophy (GA) secondary to age-related macular degeneration (AMD). Approximately 202 subjects were planned to be randomized to GT005 or the untreated control group.

Subjects entered the study had genotyping and serum complement factor I(CFI) levels assessed. Assessments were either performed at a sponsor-approved laboratory during the EXPLORE screening period or provided through participation in a previous Gyroscope sponsored study. If subjects failed to meet the eligibility criteria for EXPLORE, they were classified as screen failures for this study and could be considered for entry into another Novartis/Gyroscope sponsored study.

After providing the informed consent, subjects underwent ophthalmic and clinical assessments to determine eligibility for inclusion in the study.

Upon confirmation of eligibility, subjects in part 1 were randomized to one of two groups: low dose [2E10 vg], or high dose [2E11 vg]. Within each group, subjects were allocated to GT005 or untreated control based on a 2:1 ratio. Once part 1 enrolment was completed, and the last active subject completed screening and either was screen-failed or randomized, then Part 2 could commence. In part 2, subjects were randomized to the low dose [2E10] group or untreated control based on a 2:1 ratio. The study eye was identified for all subjects.

Subjects were stratified by GA lesion size on fundus autofluorescence (FAF) (≤10 mm2 or >10 mm2) and presence of choroidal neovascularisation (CNV) in the fellow eye (Yes or No). Randomization of study eyes in the GA lesion size upper stratum of >10 mm2 to 17.5 mm2 was capped at 20% of total subjects randomized. Once enrolment capping at 20% based on the upper GA lesion size was reached, eyes that fulfilled the cap criteria were no longer eligible, unless the subject had a CFI rare variant genotype (minor allele frequency ≤1%) previously associated with normal or low serum CFI or had an unreported CFI rare variant genotype. Of all subjects enrolled and randomized in the study, the presence of CNV in the fellow eye was capped at 25% per stratum. A permuted-block randomization method was used to obtain an approximately 2:1 ratio between GT005 and the untreated control groups for each dose group within each stratum.

Following randomization, the investigator was informed of the subject's allocated treatment (GT005 or the untreated control group) and the study eye selected. To minimize bias, all imaging endpoint assessments and grading were performed at a Central Reading Centre (CRC), in a masked fashion. For part 1, the Sponsor, subject, investigators, and study personnel performing clinical assessments remained masked to dose received for those allocated to GT005. For part 2, the Sponsor, investigators, subjects, and study personnel performing clinical assessments were unmasked to dose received, since only the low dose was administered.

Subjects randomized to GT005 underwent a single time subretinal administration of the study drug. Vitreous samples were collected during surgery. Following surgery, a prophylactic steroid regimen was prescribed.

The study consisted of a screening period lasting up to 8 weeks (or up to 12 weeks if agreed by the Sponsor Medical Monitor), followed by a 96-week study period. All subjects were assessed for the occurrence of adverse events (AEs) at each visit and underwent functional visual and retinal imaging,anatomical assessments, and biological sampling as per the schedule of assessments.

This study was conducted in compliance with Independent ethics committees (IECs) / Institutional review board (IRBs), informed consent regulations, the Declaration of Helsinki, International Council on Harmonisation (ICH) Good Clinical Practices (GCP) Guidelines, and the Food and Drug Administration (FDA) guidance.

On 24-Aug-2023, the decision was taken to terminate the study and the GT005 program. The decision was aligned with the recommendation of an independent DMC, which concluded that futility criteria had been met for the HORIZON study (GT005-03) and the overall benefit-risk ratio did not support continuation of the current development program as planned. All GT005- treated subjects, who were willing to be transferred into the long-term safety follow-up study were enrolled in the ORACLE (CPPY988A12203B / NCT05481827) study.

In both Part 1 and Part 2, patients with geographic atrophy secondary to age-related macular degeneration were enrolled. In Part 1, patients with CFI rare variant genotype and low serum CFI level and in Part 2, patients were enrolled regardless of genotypes. Efficacy results were analyzed by arm and also by part. AE and disposition data were reported per arm, but the parts were combined, according to the analysis plan.

Part 1 enrolled subjects with CFI rare variant; Part 2 enrolled subjects regardless of genotype.

There were no subjects in the high dose arm in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent
2. Age ≥55 years
3. Have a clinical diagnosis of GA secondary to AMD in the study eye, as determined by the Investigator, and a diagnosis of AMD in the contralateral eye (except if the subject is monocular)
4. Have GA lesion(s) total size between or equal to 1.25mm2 to 17.5mm2 in the study eye
5. The GA lesion(s) in the study eye must reside completely within the FAF image
6. Up to 25% of the enrolled study population are permitted to have CNV in the fellow eye, defined as either:

   1. Non-exudative/sub-clinical fellow eye CNV identified at Screening, or
   2. Known history of fellow eye CNV with either ≥2 years since diagnosis or with no active treatment required in 6 months prior to Screening
7. Have a BCVA of 24 letters (6/95 and 20/320 Snellen acuity equivalent) or better, using ETDRS charts, in the study eye
8. Part 1 Only: Subjects carrying a CFI rare variant genotype (minor allele frequency of ≤1%) previously associated with low serum CFI or subjects carrying an unreported CFI rare variant genotype that have tested to have a low serum CFI
9. Able to attend all study visits and complete the study procedures
10. Women of child-bearing potential must have a negative pregnancy test within 2 weeks prior to randomisation. A pregnancy test is not required for postmenopausal women (defined as being at least 12 consecutive months without menses) or those surgically sterilised (those having a bilateral tubal ligation/bilateral salpingectomy, bilateral tubal occlusive procedure, hysterectomy, or bilateral oophorectomy)

Exclusion Criteria:

1. Subjects who have a clinical diagnosis of Stargardt Disease or other retinal dystrophies, confirmed by the central reading centre
2. Have a history, or evidence, of CNV in the study eye
3. Presence of moderate/severe or worse non-proliferative diabetic retinopathy in the study eye
4. Have history of vitrectomy, sub-macular surgery, or macular photocoagulation in the study eye
5. History of intraocular surgery in the study eye within 12 weeks prior to Screening (Visit 1). Yttrium aluminium garnet capsulotomy is permitted if performed >10 weeks prior to Visit 1
6. Have clinically significant cataract that may require surgery during the study period in the study eye
7. Presence of moderate to severe glaucomatous optic neuropathy in the study eye; uncontrolled IOP despite the use of two or more topical agents; a history of glaucoma-filtering or valve surgery is also excluded
8. Axial myopia of greater than -8 dioptres in the study eye
9. Have any other significant ocular or non-ocular medical or psychiatric condition which, in the opinion of the Investigator, may either put the subject at risk or may influence the results of the study
10. Have a contraindication to specified protocol corticosteroid regimen
11. Have received any investigational and/or approved product(s) for the treatment of GA within the past 6 months, or 5 half-lives (whichever is longer) other than nutritional supplements such as the age-related eye disease study (AREDS) formula in the study eye or systemically
12. Have received a gene or cell therapy at any time
13. Are unwilling to use two forms of contraception (one of which being a barrier method) for 90 days post-dosing, if relevant
14. Active malignancy within the past 12 months, except for: appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or prostate cancer with a stable prostate-specific antigen (PSA) ≥12 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (32):
  - Retinal Research Institute (retina consultants of AZ), Phoenix, Arizona
  - Retina Associates of Southern California, Huntington Beach, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - Retina Consultants San Diego, Poway, California
  - VitreoRetinal Associates, P.A., Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University Retina Macula Associates PC, Lemont, Illinois
  - Midwest Eye Institute Northside, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - The Retina Care Center, Baltimore, Maryland
  - Ophthalmic Consultants of Boston (OCB), Boston, Massachusetts
  - VitreoRetinal Surgery, PLLC, Minneapolis, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Retina, Eugene, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Erie Retinal Surgery, INC, Erie, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Charles Retina Institute, Memphis, Tennessee
  - Austin Research Center for Retina, PLLC, Austin, Texas
  - Retina Consultants of Houston-TMC, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Department of Ophthalmology UW Medicine, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Australia (2):
  - The University of Melbourne - The Centre for Eye Research Australia (CERA), Melbourne E., Victoria
  - Sydney Hospital and Sydney Eye Hospital, Sydney
- France (3):
  - Centre Paradis Monticelli, Marseille, Alpes-Cote d'Azur
  - CHU Hôpital F. Mitterrand, Dijon, Bourgogne-Franche-Comté
  - CHU de Nantes - Hôtel-Dieu, Nantes, Pays de la Loire Region
- Germany (5):
  - Universitaetsklinikum Schleswig-Holstein Campus Lübeck, Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Bonn, Bonn
  - Internationale Innovative Ophthalmochirurgie, Düsseldorf
  - St. Franziskus-Hospital, Münster
  - Universitatsklinikum Tübingen, Tübingen
- Stichting Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- Oftalmika Spolka z ograniczona odpowiedzialnoscia, Bydgoszcz, Poland
- Spain (5):
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Hospital La Arruzafa, Córdoba
  - Clinica Baviera, Madrid
  - Clinica Oftalvist Valencia, Valencia
- United Kingdom (6):
  - Bristol Eye Hospital, Bristol
  - St.Paul's Eye Unit, Liverpool
  - Moorfields Eye Hospital - NHS Foundation Trust, London
  - The Retina Clinic London, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Sunderland Eye Infirmary, Sunderland

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- See also: Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, controlled study designed to evaluate the safety and efficacy of two doses of GT005 administered as a single subretinal injection in subjects with GA secondary to AMD.
  This was a study conducted in 3 treatment arms (GT005 low dose, GT005 high dose, and an untreated control group) and in 2 parts (Part 1 enrolled subjects with Complement factor I (CFI) rare variant; Part 2 enrolled subjects regardless of genotype (i.e., CFI-rare and CFI-non-rare variants));
Pre-assignment Details: The parts were determined by genotype and not treatment. Because genotype may influence disease progression, these parts were considered in the analysis of the efficacy endpoints only, but not safety, and not demographics, as pre-specified in the SAP and protocol.
Groups:
- GT005 Low Dose [2E10 vg]: GT005 Low Dose [2E10 vg]
- GT005 High Dose [2E11 vg]: GT005 High Dose [2E11 vg]
- Untreated Control: Subjects allocated to the untreated control group did not receive any treatment.
Period: Overall Study
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Started | 52 | 9 | 37
Randomized Part 1 | 10 | 9 | 14
Randomized Part 2 | 42 | 0 | 23
Randomized and Treated Part 1 | 9 | 9 | 0
Randomized and Treated Part 2 | 18 | 0 | 0
Completed | 6 | 8 | 7
Not Completed | 46 | 1 | 30
Not completed — Death | 3 | 0 | 2
Not completed — Study terminated by sponsor | 16 | 1 | 25
Not completed — Withdrawal by Subject | 4 | 0 | 3
Not completed — Sponsor instructions | 23 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) as described in the study protocol, which included all participants who were randomized to GT005 or untreated control.
  Because genotype may influence disease progression, these parts were considered in the analysis of the efficacy endpoints only, but not safety and not demographics, per the SAP and protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control | Total
Number analyzed (Participants) | 52 | 9 | 37 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.8 (7.33) | 72.7 (8.96) | 75.2 (7.07) | 75.8 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 5 | 18 | 57
  Male | 18 | 4 | 19 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 51 | 7 | 35 | 93
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline to Week 48 in Geographic Atrophy (GA) - Part 1
Description: The change from baseline to Week 48 in GA area as measured by fundus autofluorescence (FAF)
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 9 | 8 | 12
mm^2
  Part 1 Week 12 (n=9,8,12) | 0.773 (0.2151) | 0.764 (0.2159) | 0.482 (0.1848)
  Part 1 Week 24 (n=9,7,9): number analyzed (Participants) | 9 | 7 | 9
  Part 1 Week 24 (n=9,7,9) | 1.338 (0.2763) | 1.519 (0.2845) | 0.680 (0.2500)
  Part 1 Week 36 (n=6,7,10): number analyzed (Participants) | 6 | 7 | 10
  Part 1 Week 36 (n=6,7,10) | 1.800 (0.3740) | 2.044 (0.3669) | 1.132 (0.3229)
  Part 1 Week 48 (n=5,8,10): number analyzed (Participants) | 5 | 8 | 10
  Part 1 Week 48 (n=5,8,10) | 2.120 (0.3726) | 2.378 (0.3414) | 1.144 (0.3040)
Statistical Analysis 1: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.291, 90% CI 2-sided [-0.195 to 0.777], Standard Error of Mean 0.2838
Statistical Analysis 2: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.282, 90% CI 2-sided [-0.206 to 0.769], Standard Error of Mean 0.2843
Statistical Analysis 3: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.658, 90% CI 2-sided [0.017 to 1.299], Standard Error of Mean 0.3730
Statistical Analysis 4: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.840, 90% CI 2-sided [0.189 to 1.490], Standard Error of Mean 0.3791
Statistical Analysis 5: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.668, 90% CI 2-sided [-0.177 to 1.512], Standard Error of Mean 0.4954
Statistical Analysis 6: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.912, 90% CI 2-sided [0.078 to 1.746], Standard Error of Mean 0.4887
Statistical Analysis 7: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 0.976, 90% CI 2-sided [0.150 to 1.803], Standard Error of Mean 0.4813
Statistical Analysis 8: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 1.233, 90% CI 2-sided [0.445 to 2.022], Standard Error of Mean 0.4573

2. Secondary Outcome: The Change From Baseline in Geographic Atrophy (GA) at Week 72 and Week 96 - Part 1
Description: The change from baseline to Week 48 in GA area as measured by fundus autofluorescence (FAF)
Time Frame: Baseline, Weeks 72 and 96
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Least Squares Mean (Standard Error); unit: mm2
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 6 | 8 | 9
mm2
  Part 1 Week 72 (n=5,7,9): number analyzed (Participants) | 5 | 7 | 9
  Part 1 Week 72 (n=5,7,9) | 3.643 (0.9725) | 3.149 (0.9150) | 1.875 (0.8273)
  Part 1 Week 96 (n=6,8,7): number analyzed (Participants) | 6 | 8 | 7
  Part 1 Week 96 (n=6,8,7) | 4.837 (1.0712) | 4.074 (1.0305) | 2.796 (0.9240)
Statistical Analysis 1: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 1.769, 90% CI 2-sided [-0.441 to 3.979], Standard Error of Mean 1.2808
Statistical Analysis 2: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 1.274, 90% CI 2-sided [-0.863 to 3.412], Standard Error of Mean 1.2349
Statistical Analysis 3: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 2.041, 90% CI 2-sided [-0.386 to 4.468], Standard Error of Mean 1.4177
Statistical Analysis 4: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean = 1.278, 90% CI 2-sided [-1.099 to 3.655], Standard Error of Mean 1.3857

3. Secondary Outcome: Summary of Adverse Events - Parts 1 and 2 Combined
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  A TEAE is defined as any AE that develops after randomization or any AE already present that worsens following randomization. The primary summaries of AEs are based on TEAEs.
Time Frame: Adverse events are reported from randomization up to end of study, for a maximum timeframe of approximately 96 weeks.
Population: Full Analysis Set - all randomized participants. Part 1 enrolled subjects with Complement factor I (CFI) rare variant; Part 2 enrolled subjects regardless of genotype (i.e., CFI-rare and CFI-non-rare variants) . Part 1 and Part 2 are not defined in the protocol as distinct arms. Since there were no safety concerns, it was determined that there was no scientific value in reporting safety results by part / genotype, but by treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 52 | 9 | 37
Participants
  Subjects with at least one ocular adverse event for the study eye | 18 | 9 | 2
  Subjects with at least one ocular adverse event for the fellow eye | 6 | 3 | 5
  Subjects with at least one non-ocular adverse event | 13 | 8 | 14
  Subjects with at least one ocular adverse event related to study treatment for the study eye | 3 | 4 | 0
  Subjects with at least one non-ocular adverse event related to study treatment | 0 | 0 | 0
  Subjects with at least one ocular adverse event related to surgical procedure for the study eye | 12 | 7 | 0
  Subjects with at least one non-ocular adverse event related to surgical procedure | 0 | 0 | 0
  Subjects with at least one ocular adverse event related to study procedure for the study eye | 1 | 1 | 0
  Subjects with at least one non-ocular adverse event related to study procedure | 1 | 0 | 0
  Subjects with at least one ocular adverse event leading to study discontinuation for the study eye | 0 | 0 | 0
  Subjects with at least one non-ocular adverse event leading to study discontinuation | 3 | 0 | 2
  Subjects with at least one ocular adverse event of special interest for the study eye | 4 | 7 | 0
  Subjects with at least one ocular adverse event of special interest for the fellow eye | 0 | 0 | 1
  Subjects with at least one ocular serious adverse event (SAE) for the study eye | 1 | 0 | 0
  Subjects with at least one ocular serious adverse event for the fellow eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event | 5 | 2 | 4
  Subjects with at least one ocular serious adverse event related to study treatment for the study eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event related to study treatment | 0 | 0 | 0
  Subjects with at least 1 ocular SAE related to surgical procedure - study eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event related to surgical procedure | 0 | 0 | 0
  Subjects with at least one ocular serious adverse event related to study procedure for the study eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event related to study procedure | 0 | 0 | 0
  Subjects with at least 1 ocular SAE event leading to study discontinuation- study eye | 0 | 0 | 0
  Subjects with at least one non-ocular serious adverse event leading to study discontinuation | 3 | 0 | 2
  Deaths | 3 | 0 | 2

4. Secondary Outcome: Ocular Adverse Events by Primary System Organ Class and Preferred Term for the Study Eye - Parts 1 and 2 Combined
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject.
  A TEAE is defined as any AE that develops after randomization or any AE already present that worsens following randomization. The primary summaries of AEs are based on TEAEs.
  System organ classes are sorted alphabetically, and preferred terms are sorted by decreasing overall frequency within system organ class.
Time Frame: Adverse events are reported from randomization up to end of study, for a maximum timeframe of approximately 96 weeks.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 52 | 9 | 37
Participants
  Subjects with at least one event | 18 | 9 | 2
  Eye disorders | 15 | 9 | 2
  -Retinal pigmentation | 3 | 6 | 0
  -Conjunctival haemorrhage | 6 | 1 | 0
  -Cataract | 3 | 2 | 1
  -Cataract nuclear | 2 | 1 | 0
  -Eye pain | 1 | 2 | 0
  -Retinal haemorrhage | 2 | 1 | 0
  -Anterior chamber cell | 1 | 1 | 0
  -Blepharitis | 2 | 0 | 0
  -Conjunctivitis allergic | 1 | 1 | 0
  -Anterior chamber flare | 0 | 1 | 0
  -Choroidal detachment | 0 | 1 | 0
  -Conjunctival hyperaemia | 1 | 0 | 0
  -Dry eye | 1 | 0 | 0
  -Eye pruritus | 0 | 0 | 1
  -Hypotony maculopathy | 0 | 1 | 0
  -Iridocyclitis | 0 | 1 | 0
  -Iritis | 1 | 0 | 0
  -Keratitis | 1 | 0 | 0
  -Lacrimation increased | 0 | 1 | 0
  -Macular hole | 1 | 0 | 0
  -Meibomian gland dysfunction | 1 | 0 | 0
  -Metamorphopsia | 1 | 0 | 0
  -Ocular hypertension | 1 | 0 | 0
  -Open angle glaucoma | 0 | 1 | 0
  -Photophobia | 0 | 1 | 0
  -Photopsia | 1 | 0 | 0
  -Posterior capsule opacification | 0 | 0 | 1
  -Punctate keratitis | 1 | 0 | 0
  -Retinal depigmentation | 1 | 0 | 0
  -Visual acuity reduced | 1 | 0 | 0
  -Visual impairment | 1 | 0 | 0
  -Visual snow syndrome | 1 | 0 | 0
  -Vitreous floaters | 1 | 0 | 0
  -Vitreous haemorrhage | 1 | 0 | 0
  Injury, poisoning and procedural complications | 4 | 1 | 0
  -Post procedural discomfort | 2 | 0 | 0
  -Procedural pain | 1 | 1 | 0
  -Suture related complication | 1 | 1 | 0
  Investigations | 4 | 3 | 0
  -Intraocular pressure increased | 4 | 3 | 0
  Skin and subcutaneous tissue disorders | 1 | 0 | 0
  -Telangiectasia | 1 | 0 | 0

5. Secondary Outcome: Non-ocular Adverse Events - Summary - Parts 1 and 2 Combined
Description: as for outcome 3
Time Frame: Adverse events are reported from randomization up to end of study, for a maximum timeframe of approximately 96 weeks.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 52 | 9 | 37
Participants | 13 | 8 | 14

6. Secondary Outcome: Change in GA Morphology From Baseline to Week 96 on Colour Fundus Photography (CFP) - Number of Participants With Increase in Fundus Autofluorescence (FAF) - Part 1
Description: Change in GA morphology on multimodal imaging through Week 96.
  FAF images at Week 5 were introduced via a protocol amendment after most participants had already completed Week 5; therefore, only a minimal number of patients had FAF images taken at Week 5 for Part 1.
Time Frame: Baseline, Weeks 5,12,24,36,48,72,96
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 9 | 8 | 12
Participants
  Part 1 Week 5 (n= 0,2,0): number analyzed (Participants) | 0 | 2 | 0
  Part 1 Week 5 (n= 0,2,0) |  | 2 |
  Part 1 Week 12 (n=9,8,12) | 8 | 8 | 11
  Part 1 Week 24 (n=9,7,10): number analyzed (Participants) | 9 | 7 | 10
  Part 1 Week 24 (n=9,7,10) | 8 | 7 | 10
  Part 1 Week 36 (n=6,7,10): number analyzed (Participants) | 6 | 7 | 10
  Part 1 Week 36 (n=6,7,10) | 5 | 7 | 10
  Part 1 Week 48 (n=5,8,10): number analyzed (Participants) | 5 | 8 | 10
  Part 1 Week 48 (n=5,8,10) | 5 | 8 | 10
  Part 1 Week 72 (n=5,8,9): number analyzed (Participants) | 5 | 8 | 9
  Part 1 Week 72 (n=5,8,9) | 5 | 8 | 9
  Part 1 Week 96 (n=6,8,7): number analyzed (Participants) | 6 | 8 | 7
  Part 1 Week 96 (n=6,8,7) | 6 | 8 | 7

7. Secondary Outcome: Change From Baseline to Week 48 in GA Morphology on Colour Fundus Photography (CFP) - Number of Participants With Increase in Fundus Autofluorescence - Part 2
Description: Change in GA morphology on multimodal imaging through Week 48.
  For the untreated control group, there were no protocol-specified visits for Weeks 5 and 8.
  The untreated control participants were immediately discontinued from the study when the study was early terminated; therefore Week 36 and 48 data in part 2 were not applicable for these the untreated control group.
Time Frame: Baseline, Weeks 5,12,24,36,48
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 17 | 0 | 20
Participants
  Part 2 Week 5 (n= 16,0, 0): number analyzed (Participants) | 16 | 0 | 0
  Part 2 Week 5 (n= 16,0, 0) | 16 |  |
  Part 2 Week 12 (n=17,0,20) | 17 |  | 20
  Part 2 Week 24 (n=17,0,11): number analyzed (Participants) | 17 | 0 | 11
  Part 2 Week 24 (n=17,0,11) | 16 |  | 11
  Part 2 Week 36 (n=14,0,0): number analyzed (Participants) | 14 | 0 | 0
  Part 2 Week 36 (n=14,0,0) | 13 |  |
  Part 2 Week 48 (n=5,0,0): number analyzed (Participants) | 5 | 0 | 0
  Part 2 Week 48 (n=5,0,0) | 5 |  |

8. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) Score From Baseline Through Week 96 Via the Early Treatment for Diabetic Retinopathy (ETDRS) Chart - Part 1
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
  For the untreated control group, there were no protocol-specified visits for Weeks 1, 5 and 8.
Time Frame: Baseline, Weeks 1, 5, 8, 12, 24, 36, 48, 72 and 96
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Least Squares Mean (Standard Error); unit: Letters read
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 9 | 9 | 12
Letters read
  Part 1 - Week 1 (n=9,9,0): number analyzed (Participants) | 9 | 9 | 0
  Part 1 - Week 1 (n=9,9,0) | -4.7 (4.04) | -5.2 (4.27) |
  Part 1 - Week 5 (n=8,9,0): number analyzed (Participants) | 8 | 9 | 0
  Part 1 - Week 5 (n=8,9,0) | -1.7 (4.08) | -7.6 (4.26) |
  Part 1 - Week 8 (n=9,9,0): number analyzed (Participants) | 9 | 9 | 0
  Part 1 - Week 8 (n=9,9,0) | -1.6 (4.03) | -4.5 (4.23) |
  Part 1 - Week 12 (N=9,9,12) | -2.3 (4.03) | -7.5 (4.18) | -1.2 (3.81)
  Part 1 - Week 24 (n=9,9,10): number analyzed (Participants) | 9 | 9 | 10
  Part 1 - Week 24 (n=9,9,10) | -5.6 (4.03) | -12.0 (4.18) | -0.4 (3.87)
  Part 1 - Week 36 (n=8,8,10): number analyzed (Participants) | 8 | 8 | 10
  Part 1 - Week 36 (n=8,8,10) | -10.0 (4.10) | -12.9 (4.28) | -1.0 (3.89)
  Part 1 - Week 48 (n=5,8,10): number analyzed (Participants) | 5 | 8 | 10
  Part 1 - Week 48 (n=5,8,10) | -8.6 (4.52) | -13.3 (4.32) | -5.7 (3.91)
  Part 1 - Week 72 (n=5,8,10): number analyzed (Participants) | 5 | 8 | 10
  Part 1 - Week 72 (n=5,8,10) | -6.3 (4.56) | -9.6 (4.34) | -8.9 (3.94)
  Part 1 - Week 96 (n=6,8,7): number analyzed (Participants) | 6 | 8 | 7
  Part 1 - Week 96 (n=6,8,7) | -6.5 (4.50) | -11.0 (4.33) | -7.9 (4.30)
Statistical Analysis 1: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -1.1, 90% CI 2-sided [-10.3 to 8.1], Standard Error of Mean 5.49
Statistical Analysis 2: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 12; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -6.3, 90% CI 2-sided [-16.3 to 3.7], Standard Error of Mean 5.96
Statistical Analysis 3: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -5.2, 90% CI 2-sided [-14.5 to 4.1], Standard Error of Mean 5.54
Statistical Analysis 4: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 24; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -11.7, 90% CI 2-sided [-21.7 to -1.6], Standard Error of Mean 6.00
Statistical Analysis 5: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -9.0, 90% CI 2-sided [-18.4 to 0.5], Standard Error of Mean 5.63
Statistical Analysis 6: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 36; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -11.9, 90% CI 2-sided [-22.1 to -1.7], Standard Error of Mean 6.08
Statistical Analysis 7: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -2.9, 90% CI 2-sided [-12.7 to 6.9], Standard Error of Mean 5.88
Statistical Analysis 8: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 48; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -7.6, 90% CI 2-sided [-17.9 to 2.7], Standard Error of Mean 6.14
Statistical Analysis 9: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 2.6, 90% CI 2-sided [-7.4 to 12.5], Standard Error of Mean 5.96
Statistical Analysis 10: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 72; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -0.7, 90% CI 2-sided [-11.1 to 9.6], Standard Error of Mean 6.18
Statistical Analysis 11: Comparison: GT005 Low Dose [2E10 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean Difference = 1.4, 90% CI 2-sided [-8.7 to 11.5], Standard Error of Mean 6.07
Statistical Analysis 12: Comparison: GT005 High Dose [2E11 vg] vs Untreated Control; Week 96; Test type: Superiority; mixed model repeated measures; LS Mean Difference = -3.0, 90% CI 2-sided [-13.8 to 7.8], Standard Error of Mean 6.47

9. Secondary Outcome: Change in Low Luminance Difference (LLD) Letter Count From Baseline at Weeks 12, 24, 36, 48, 72 and 96, Via Early Treatment for Diabetic Retinopathy (ETDRS) Chart - Part 1
Description: LLD was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  The test was to be performed after BCVA testing, prior to pupil dilation, and distance refraction was to be carried out before Low Luminance Visual Acuity (LLVA) was measured.
  LLVA was to be measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the subject read the normally illuminated ETDRS chart. The LLD was calculated as the difference between BCVA and LLVA.
  Initially, letters were to be read at a distance of 4 metres from the chart. If <20 letters were read at 4 metres, testing at 1 metre should have been performed. LLD was to be reported as number of letters read correctly by the subject.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72 and 96
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 9 | 9 | 12
Letters read
  Part 1 - Week 12 (N=9,9,12) | 2.0 (9.06) | 2.4 (22.49) | -2.0 (7.21)
  Part 1 - Week 24 (n=9,9,10): number analyzed (Participants) | 9 | 9 | 10
  Part 1 - Week 24 (n=9,9,10) | 2.1 (8.40) | 2.9 (24.81) | -2.9 (7.68)
  Part 1 - Week 36 (n=8,8,10): number analyzed (Participants) | 8 | 8 | 10
  Part 1 - Week 36 (n=8,8,10) | 2.3 (15.65) | -7.5 (19.41) | -4.0 (12.51)
  Part 1 - Week 48 (n=5,8,10): number analyzed (Participants) | 5 | 8 | 10
  Part 1 - Week 48 (n=5,8,10) | 3.0 (6.96) | 1.8 (26.25) | -6.2 (19.99)
  Part 1 - Week 72 (n=5,8,10): number analyzed (Participants) | 5 | 8 | 10
  Part 1 - Week 72 (n=5,8,10) | 4.4 (7.57) | 3.1 (32.24) | -6.6 (21.15)
  Part 1 - Week 96 (n=6,8,6): number analyzed (Participants) | 6 | 8 | 6
  Part 1 - Week 96 (n=6,8,6) | 5.2 (8.47) | 1.5 (29.17) | -10.5 (27.41)

10. Secondary Outcome: Change in Low Luminance Difference (LLD) Letter Count From Baseline at Weeks 12, 24, 36, and 48, Via Early Treatment for Diabetic Retinopathy (ETDRS) Chart - Part 2
Description: as for outcome 9
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact. The untreated control participants were immediately discontinued from the study when the study was early terminated; therefore Week 36 and 48 data in part 2 were not applicable for these the untreated control group.
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 18 | 0 | 20
Letters read
  Part 2 - Week 12 (N=18,0,20) | 0.7 (10.83) |  | -1.4 (11.76)
  Part 2 - Week 24 (n=17,0,10): number analyzed (Participants) | 17 | 0 | 10
  Part 2 - Week 24 (n=17,0,10) | 2.6 (9.98) |  | -1.6 (20.13)
  Part 2 - Week 36 (n=14,0,0): number analyzed (Participants) | 14 | 0 | 0
  Part 2 - Week 36 (n=14,0,0) | 4.6 (11.77) |  |
  Part 2 - Week 48 (n=5,0,0): number analyzed (Participants) | 5 | 0 | 0
  Part 2 - Week 48 (n=5,0,0) | -2.8 (4.32) |  |

11. Secondary Outcome: Change From Baseline at Weeks 24, 36, 48, 72 and 96 in Reading Performance, Measured as the Maximum Reading Speed (Words Per Minute), as Assessed by Minnesota Low-vision Reading Test (MNRead) Chart - Part 1
Description: The maximum reading speed (MRS) represents the highest reading speed an individual can achieve when print size is not a limiting factor. Essentially, it measures how quickly a person can read text when the print is large enough to be easily readable.
  A higher count represents better visual functioning.
Time Frame: Baseline, Weeks 24, 36, 48, 72 and 96
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Words read per minute
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 9 | 8 | 9
Words read per minute
  Part 1 - Week 24 (n=9,8,9) | 20.384 (74.7769) | -36.154 (40.3322) | -7.837 (21.8918)
  Part 1 - Week 36 (n=7,7,8): number analyzed (Participants) | 7 | 7 | 8
  Part 1 - Week 36 (n=7,7,8) | -15.048 (33.0479) | -34.653 (27.2693) | -15.245 (22.0983)
  Part 1 - Week 48 (n=4,7,9): number analyzed (Participants) | 4 | 7 | 9
  Part 1 - Week 48 (n=4,7,9) | 10.397 (11.8698) | -36.285 (40.0938) | -6.837 (31.6162)
  Part 1 - Week 72 (n=5,7,9): number analyzed (Participants) | 5 | 7 | 9
  Part 1 - Week 72 (n=5,7,9) | -20.796 (42.2571) | -44.913 (46.7594) | -15.429 (30.1012)
  Part 1 - Week 96 (n=6,5,5): number analyzed (Participants) | 6 | 5 | 5
  Part 1 - Week 96 (n=6,5,5) | 10.802 (32.1161) | -32.266 (36.9172) | -21.602 (26.0643)

12. Secondary Outcome: Change From Baseline at Weeks 24, 36 and 48 in Reading Performance, Measured as the Maximum Reading Speed (Words Per Minute), as Assessed by Minnesota Low-vision Reading Test (MNRead) Chart - Part 2
Description: A higher count represents better visual functioning.
  The untreated control participants were immediately discontinued from the study when the study was early terminated; therefore Week 36 and 48 data in part 2 were not applicable for these the untreated control group.
Time Frame: Baseline, Weeks 24, 36 and 48
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Words read per minute
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 16 | 0 | 10
Words read per minute
  Part 2 - Week 24 (n=16,0,10) | 15.581 (78.2848) |  | -30.707 (27.3225)
  Part 2 - Week 36 (n=14,0,0): number analyzed (Participants) | 14 | 0 | 0
  Part 2 - Week 36 (n=14,0,0) | 9.812 (94.4255) |  |
  Part 2 - Week 48 (n=5,0,0): number analyzed (Participants) | 5 | 0 | 0
  Part 2 - Week 48 (n=5,0,0) | -28.111 (38.6209) |  |

13. Secondary Outcome: Change From Baseline at Weeks 24, 36, 48, 72 and 96 in Functional Reading Independence (FRI) Index - Part 1
Description: The FRI index is a patient-reported outcome measure developed specifically for use in GA patients. The FRI index evaluates the level of independence subjects have in performing everyday activities that require reading, such as writing a cheque or reading a prescription.
  Scores derived from the index range from 1 (unable to do) to 4 (total independence).
  A higher score represents better visual functioning.
Time Frame: Baseline, Weeks 24, 36, 48, 72 and 96
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 9 | 8 | 10
Scores on a scale
  Part 1 - Week 24 (n=9,8,10) | 0.7 (3.57) | -1.3 (2.55) | -0.3 (4.06)
  Part 1 - Week 36 (n=8,5,10): number analyzed (Participants) | 8 | 5 | 10
  Part 1 - Week 36 (n=8,5,10) | -1.0 (4.24) | 2.6 (4.10) | -0.6 (4.72)
  Part 1 - Week 48 (n=6,7,10): number analyzed (Participants) | 6 | 7 | 10
  Part 1 - Week 48 (n=6,7,10) | 0.5 (2.43) | -0.1 (7.69) | -3.4 (4.38)
  Part 1 - Week 72 (n=5,7,10): number analyzed (Participants) | 5 | 7 | 10
  Part 1 - Week 72 (n=5,7,10) | -3.8 (4.60) | 0.4 (3.41) | -1.3 (4.35)
  Part 1 - Week 96 (n=6,6,7): number analyzed (Participants) | 6 | 6 | 7
  Part 1 - Week 96 (n=6,6,7) | -2.7 (5.79) | -2.0 (3.29) | -0.7 (5.53)

14. Secondary Outcome: Change From Baseline at Weeks 24, 36 and 48 in Functional Reading Independence (FRI) Index - Part 2
Description: The FRI index is a patient-reported outcome measure developed specifically for use in GA patients. The FRI index evaluates the level of independence subjects have in performing everyday activities that require reading, such as writing a cheque or reading a prescription.
  Scores derived from the index range from 1 (unable to do) to 4 (total independence).
  A higher score represents better visual functioning.
  The untreated control participants were immediately discontinued from the study when the study was early terminated; therefore Week 36 and 48 data in part 2 were not applicable for these the untreated control group.
Time Frame: Baseline, Weeks 24, 36 and 48
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 17 | 0 | 9
Scores on a scale
  Part 2 - Week 24 (n=17,0,9) | -0.4 (2.83) |  | 0.4 (6.86)
  Part 2 - Week 36 (n=14,0,0): number analyzed (Participants) | 14 | 0 | 0
  Part 2 - Week 36 (n=14,0,0) | -1.7 (3.83) |  |
  Part 2 - Week 48 (n=5,0,0): number analyzed (Participants) | 5 | 0 | 0
  Part 2 - Week 48 (n=5,0,0) | 0.4 (5.13) |  |

15. Secondary Outcome: Change From Baseline at Weeks 24, 36, 48, 72 and 96 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Composite Score - Part 1
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures the influence of visual disability and visual symptoms on general health domains.
  The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better visual functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. A composite score is derived based on the average of the 11 subscales.
Time Frame: Baseline, Weeks 24, 36, 48, 72 and 96
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 9 | 9 | 10
Scores on a Scale
  Part 1 - Week 24 (n=9,9,10) | -2.312 (5.7079) | -3.755 (7.4470) | -7.304 (12.5136)
  Part 1 - Week 36 (n=8,6,10): number analyzed (Participants) | 8 | 6 | 10
  Part 1 - Week 36 (n=8,6,10) | -4.400 (11.1307) | 1.960 (9.0113) | -4.706 (11.8617)
  Part 1 - Week 48 (n=6,8,10): number analyzed (Participants) | 6 | 8 | 10
  Part 1 - Week 48 (n=6,8,10) | -6.439 (24.2128) | -6.810 (11.5980) | -4.091 (15.3598)
  Part 1 - Week 72 (n=5,8,10): number analyzed (Participants) | 5 | 8 | 10
  Part 1 - Week 72 (n=5,8,10) | -8.698 (22.1289) | -3.332 (8.1470) | -3.826 (11.0029)
  Part 1 - Week 96 (n=6,7,7): number analyzed (Participants) | 6 | 7 | 7
  Part 1 - Week 96 (n=6,7,7) | -10.352 (23.9470) | 0.171 (11.3543) | -10.700 (11.6900)

16. Secondary Outcome: Change From Baseline at Weeks 24, 36 and 48 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Composite Score - Part 2
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures the influence of visual disability and visual symptoms on general health domains.
  The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better visual functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. A composite score is derived based on the average of the 11 subscales.
  The untreated control participants were immediately discontinued from the study when the study was early terminated; therefore Week 36 and 48 data in part 2 were not applicable for these the untreated control group.
Time Frame: Baseline, Weeks 24, 36, and 48
Population: Full Analysis Set - for randomized participants with a valid measurement without a protocol deviation with impact.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control
Number analyzed (Participants) | 17 | 0 | 8
Scores on a Scale
  Part 2 - Week 24 (n=17,0,8) | -4.034 (6.8881) |  | -3.070 (7.4251)
  Part 2 - Week 36 (n=14,0,0): number analyzed (Participants) | 14 | 0 | 0
  Part 2 - Week 36 (n=14,0,0) | -2.733 (7.9219) |  |
  Part 2 - Week 48 (n=5,0,0): number analyzed (Participants) | 5 | 0 | 0
  Part 2 - Week 48 (n=5,0,0) | -0.530 (6.9722) |  |

ADVERSE EVENTS:
Time Frame: Adverse events are reported from randomization up to end of study, for a maximum timeframe of approximately 96 weeks.
Description: Full Analysis Set - all randomized participants. Part 1 enrolled subjects with Complement factor I (CFI) rare variant; Part 2 enrolled subjects regardless of genotype (i.e., CFI-rare and CFI-non-rare variants) . Part 1 and Part 2 are not defined in the protocol as distinct arms. Since there were no safety concerns, it was determined that there was no scientific value in reporting safety results by part / genotype, but by treatment.
Groups:
- Overall: Overall
Arm/Group | GT005 Low Dose [2E10 vg] | GT005 High Dose [2E11 vg] | Untreated Control | Overall
All-Cause Mortality (participants affected / at risk) | 3/52 | 0/9 | 2/37 | 5/98
Serious Adverse Events (participants affected / at risk) | 5/52 | 2/9 | 4/37 | 11/98
Other Adverse Events (participants affected / at risk) | 19/52 | 9/9 | 16/37 | 44/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GT005 Low Dose [2E10 vg] (N=52) | GT005 High Dose [2E11 vg] (N=9) | Untreated Control (N=37) | Overall (N=98)
Visual acuity reduced - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GT005 Low Dose [2E10 vg] (N=52) | GT005 High Dose [2E11 vg] (N=9) | Untreated Control (N=37) | Overall (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Anterior chamber cell - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Anterior chamber flare - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Blepharitis - Fellow eye (Eye disorders) | 2 | 0 | 0 | 2
Blepharitis - Study eye (Eye disorders) | 2 | 0 | 0 | 2
Cataract - Fellow eye (Eye disorders) | 0 | 1 | 2 | 3
Cataract - Study eye (Eye disorders) | 3 | 2 | 1 | 6
Cataract nuclear - Study eye (Eye disorders) | 2 | 1 | 0 | 3
Choroidal detachment - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Choroidal neovascularisation - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Conjunctival haemorrhage - Study eye (Eye disorders) | 6 | 1 | 0 | 7
Conjunctival hyperaemia - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Conjunctivitis allergic - Fellow eye (Eye disorders) | 1 | 1 | 0 | 2
Conjunctivitis allergic - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Dry eye - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Dry eye - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Eye pain - Study eye (Eye disorders) | 1 | 2 | 0 | 3
Eye pruritus - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Eye pruritus - Study eye (Eye disorders) | 0 | 0 | 1 | 1
Hypotony maculopathy - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Iridocyclitis - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Iritis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Keratitis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Lacrimation increased - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Macular hole - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Meibomian gland dysfunction - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Meibomian gland dysfunction - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Metamorphopsia - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Ocular hypertension - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Open angle glaucoma - Fellow eye (Eye disorders) | 0 | 1 | 0 | 1
Open angle glaucoma - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Photophobia - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Photopsia - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Photopsia - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Posterior capsule opacification - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Posterior capsule opacification - Study eye (Eye disorders) | 0 | 0 | 1 | 1
Punctate keratitis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Retinal degeneration - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Retinal depigmentation - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Retinal haemorrhage - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Retinal haemorrhage - Study eye (Eye disorders) | 2 | 1 | 0 | 3
Retinal oedema - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Retinal pigmentation - Study eye (Eye disorders) | 3 | 6 | 0 | 9
Retinal tear - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Visual impairment - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Visual impairment - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Visual snow syndrome - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Vitreous detachment - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Vitreous floaters - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Vitreous floaters - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Vitreous haemorrhage - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 1
Drug intolerance (General disorders) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 3 | 2 | 1 | 6
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 1 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural discomfort - Study eye (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Procedural pain - Study eye (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Suture related complication - Study eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 1 | 2
Intraocular pressure increased - Study eye (Investigations) | 4 | 3 | 0 | 7
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urethral polyp (Renal and urinary disorders) | 0 | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Telangiectasia - Fellow eye (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Telangiectasia - Study eye (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT04437368/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT04437368/SAP_001.pdf